CLINICAL TRIAL: NCT06675981
Title: Placebo Response of Different Types of Sham Acupuncture for Knee Osteoarthritis
Acronym: PSAKOA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Sun Xin, professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 82305045; 82305045 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
Keywords: Sham acupuncture; Randomized controlled trial; Blinding effect; Placebo acupuncture
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Real Acupuncture (Experimental): Acupuncture at nine acupoints. Patients received 6 sessions of acupuncture (three sessions per week or every other day) for two consecutive weeks
  Interventions: Other: Real Acupuncture
- Non-acupuncture at real-acupoint (Sham Comparator): The acupuncture simulation device will be used to perform acupuncture at the same acupoints as those of the real acupuncture group.
  Interventions: Other: Non-acupuncture at real-acupoint
- Shallow acupuncture at real-acupoint (Sham Comparator): At the same acupoint in the acupuncture group, the subcutaneous puncture is only 1-2 mm, no manipulation will be applied
  Interventions: Other: Shallow acupuncture at real-acupoint
- Shallow acupuncture at non-meridian and non-acupoint (Sham Comparator): At non-meridian and non-acupoint, the subcutaneous puncture is only 1-2 mm, no manipulation will be applied
  Interventions: Other: Shallow acupuncture at non-meridian and non-acupoint
- Waiting-list group (No Intervention): No acupuncture treatment will be given during the study period.

INTERVENTIONS:
Other: Real Acupuncture — Patients received 6 sessions of acupuncture (three sessions per week or every other day) for two consecutive weeks
  Arms: Real Acupuncture
Other: Non-acupuncture at real-acupoint — The acupuncture simulation device will be used to perform acupuncture at the same acupoints as those of the real acupuncture group.
  Arms: Non-acupuncture at real-acupoint
Other: Shallow acupuncture at real-acupoint — At the same acupoint in the acupuncture group, the subcutaneous puncture is only 1-2 mm, no manipulation will be applied
  Arms: Shallow acupuncture at real-acupoint
Other: Shallow acupuncture at non-meridian and non-acupoint — At non-meridian and non-acupoint, the subcutaneous puncture is only 1-2 mm, no manipulation will be applied
  Arms: Shallow acupuncture at non-meridian and non-acupoint

SUMMARY:
This study aims to conduct a randomized controlled trial to investigate the difference in clinical efficacy and blinding effect between real acupuncture and various sham acupuncture techniques.

DETAILED DESCRIPTION:
This study aimed to recruit 150 patients with knee osteoarthritis from the hospital outpatient department. Random coding was generated using a computer network-based random system, and the subjects will be divided into five groups: real acupuncture, non-acupuncture at real-acupoint, shallow acupuncture at real-acupoint, shallow acupuncture at non-meridian and non-acupoint, and waiting treatment group in a 1:1:1:1 ratio. Acupuncture sessions were conducted three times a week for two weeks. Patients in the waiting treatment group did not receive acupuncture therapy during the study period but received acupuncture treatment after the trial. Outcome measures included Western Ontario and McMaster Universities Osteoarthritis index (WOMAC) score, Visual Analogue Pain (VAS) score, Massachusetts General Hospital Acupuncture Sensation Scale (MASS) needle sensation score, and blind evaluation scale. Data collection occurred at baseline, one week, and two weeks.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of knee osteoarthritis.
* Age over 40 years old.

Exclusion criteria:

* Tuberculosis, tumors, rheumatism of the knee joint, and rheumatoid arthritis.
* Sprain or trauma in the lower limb.
* Mental disorders.
* Severe cardiovascular disease, liver or kidney impairment, immunodeficiency, diabetes mellitus, blood disorder or skin disease.
* Pregnancy or lactation.
* Use of physiotherapy for osteoarthritis knee pain in the past month; use of intra-articular injection of glucocorticoid or viscosupplementation in the past 6 months; received knee-replacement surgery; and positive floating patella test.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis index (WOMAC) | 2 week
  The WOMAC, a disease-specific scale with high reliability and validity, has been translated into different languages and used widely in clinical trials for KOA. The Chinese version of WOMAC contains 24 items that measure pain (5 items, scored 0-50), stiffness (2 items, scored 0-20) and physical function (17 items, scored 0-170), with a total score ranging from 0 to 240

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | 2 week
  The Visual Analogue Scale (VAS) measures pain on a scale of 0 to 10, with a higher score indicating more severe symptoms.
Blind Assessment Scale | 2 week
  The patients in the real acupuncture and sham acupuncture groups will be asked, "Do you think you are receiving real acupuncture treatment?" The patients' response options were "yes, no, and not sure."
Massachusetts General Hospital Acupuncture Sensation Scale (MASS) | 2 week
  The scale consists of 13 items and measures the body sensation experienced during acupuncture, including sensations such as acid, numbness, distension, pain, and heat. Each of the 13 entries utilizes a Visual Analogue Scale (VAS) with a range from 0cm (indicating no needle sensation) to 10cm (representing strong to unbearable needle sensation).

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, Doctor, Study Chair — West China Hospital
Locations (2):
- China (2):
  - Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine, Nanchang, Jiangxi
  - Affiliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers with the agreement of the Coordinating Committee and the Ethics Committee.